CLINICAL TRIAL: NCT05493605
Title: Cardiac Involvement in Wilson's Disease
Acronym: WIL-HEART
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: APS_2021_9
Record Dates: First submitted 2022-07-21; First posted 2022-08-09 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Wilson's Disease
MeSH Terms: conditions — Hepatolenticular Degeneration

STUDY DESIGN:
Intervention Model Description: All patients with confirmed Wilson Disease presenting for consultation or hospitalization for their follow-up or at the time of diagnosis will be offered to participate in the study.
  Patients who have already benefited from a cardiac assessment with installation of an implantable Holter ECG as part of the treatment may be included retrospectively
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cases (Other): The intervention consists in setting up a morphological and rhythmological cardiological follow-up patients with confirmed Wilson disease. It will require the wearing of a long Holter duration (21 days) and for some patients the installation of an implantable cardiac monitor.The long-time ECG holter is used to record heart rhythm for 21 days and detect possible arrhythmias (accelerations of the heart) or conduction disorders (slowdowns of the heart).
  Interventions: Procedure: Delivery of a long-term Holter 21 days Or placement of an implantable holter from the outset so syncope

INTERVENTIONS:
Procedure: Delivery of a long-term Holter 21 days Or placement of an implantable holter from the outset so syncope — The intervention consists of setting up a morphological and rhythmological cardiological follow-up of patients with confirmed Wilson's disease. It will require the wearing of a long-term Holter (21 days) and for some patients the installation of an implantable cardiac monitor.

SUMMARY:
Heart damage by copper accumulation has been reported in Wilson's Disease. However, the disease epidemiology is still poorly understood. A number of studies on pediatric populations have not shown any significant cardiac involvement apart from early dysautonomia. This could suggest that the clinical manifestations related to the copper accumulation in the heart appears with the duration of the disease. Case-control studies on adult populations have highlighted various electrocardiographic (ECG) abnormalities more frequent in patients with Wilson's Disease than in healthy volunteers, but all these studies involved small number of patients (maximum 60). The hypothesis is that there is cardiac involvement in Wilson's Disease, requiring screening, follow-up and appropriate support.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient with Wilson's disease confirmed by a Leipzig score ≥ 4
* Express consent to participate in the study by the patient or legal guardian in the case of patients under guardianship or by the patient assisted by his curator in the case of patients under guardianship
* Member of or beneficiary of a Social Security scheme

Exclusion Criteria:

* Absolute or relative contraindication to MRI or contrast media
* Pregnant, parturient or breast-feeding women: a urine pregnancy test will be carried out in women of childbearing age
* Patient with hepatic decompensation (Child-Pugh score stage C)
* Patient in neuro-psychiatric decompensation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-03-02 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Contrast-enhanced cardiac MRI - Day 0 | Day 0
  Percentage of patients with abnormal contrast-enhanced cardiac MRI results
Contrast-enhanced cardiac MRI - Day 0 | Day 0
  Description of abnormalities (frequency and percentage)
Transthoracic echocardiography - Day 0 | Day 0
  Percentage of patients with abnormal transthoracic echocardiography results
Transthoracic echocardiography - Day 0 | Day 0
  Description of abnormalities (frequency and percentage)
Chest computed tomography scan without contrast - Day 0 | Day 0
  Percentage of patients with abnormal coronary artery calcium score
  Calcium score : The higher the coronary calcium score, the greater the cardiovascular risk. A score of 0 (min) means that no calcium is seen in the heart. A score greater than 300 is a sign of very high to severe disease.
Electrocardiogram - Day 0 | Day 0
  Percentage of patients with abnormal electrocardiogram results
Electrocardiogram - Day 0 | Day 0
  Description of abnormalities (frequency and percentage)
Clinical examination - Day 0 | Day 0
  Percentage of patients with abnormal clinical examination
Clinical examination - Day 0 | Day 0
  Description of abnormalities (frequency and percentage)
Blood and urine tests - Day 0 | Day 0
  Percentage of patients with abnormal blood and urine tests results Blood tests performed : lipid profile, glycosylated hemoglobin (HbA1C), cardiac enzymes (troponin C, NT-proBNP), ultra-sensitive C-reactive protein, sodium level, potassium level, urea and creatinine clearance, TSH, fibrinogen Urine test performed : proteinuria
Blood and urine tests - Day 0 | Day 0
  Description of abnormalities (frequency and percentage) Blood tests performed : lipid profile, glycosylated hemoglobin (HbA1C), cardiac enzymes (troponin C, NT-proBNP), ultra-sensitive C-reactive protein, sodium level, potassium level, urea and creatinine clearance, TSH, fibrinogen Urine test performed : proteinuria
Lying and standing blood pressure tests - Day 0 | Day 0
  Percentage of patients with abnormal blood pressure tests results
Lying and standing blood pressure tests - Day 0 | Day 0
  Description of abnormalities (frequency and percentage)
Implantable loop recorder or ECG holter recorder- Day 21 | Day 21
  Percentage of patients with abnormal implantable loop record (or ECG holter record) The device will record from Day 0 to Day 21 Implantable loop recorder assessment will be only performed on patients with syncope.
Implantable loop recorder or ECG holter recorder- Day 21 | Day 21
  Description of abnormalities (frequency and percentage) The device will record from Day 0 to Day 21 Implantable loop recorder assessment will be only performed on patients with syncope.
Transthoracic echocardiography - Year 3 | Year 3
  Percentage of patients with abnormal transthoracic echocardiography results
Transthoracic echocardiography - Year 3 | Year 3
  Description of abnormalities (frequency and percentage)
Contrast-enhanced cardiac MRI - Year 3 | Year 3
  Percentage of patients with abnormal contrast-enhanced cardiac MRI results
Contrast-enhanced cardiac MRI - Year 3 | Year 3
  Description of abnormalities (frequency and percentage)
Chest computed tomography scan without contrast - Year 3 | Year 3
  Percentage of patients with abnormal coronary artery calcium score
  Calcium score : The higher the coronary calcium score, the greater the cardiovascular risk. A score of 0 (min) means that no calcium is seen in the heart. A score greater than 300 is a sign of very high to severe disease.
Electrocardiogram - Year 3 | Year 3
  Percentage of patients with abnormal electrocardiogram results
Electrocardiogram - Year 3 | Year 3
  Description of abnormalities (frequency and percentage)
Clinical examination - Year 3 | Year 3
  Percentage of patients with abnormal clinical examination
Clinical examination - Year 3 | Year 3
  Description of abnormalities (frequency and percentage)
Blood and urine tests - Year 3 | Year 3
  Percentage of patients with abnormal blood or urine tests results Blood tests performed : lipid profile, glycosylated hemoglobin (HbA1C), cardiac enzymes (troponin C, NT-proBNP), ultra-sensitive C-reactive protein, sodium level, potassium level, urea and creatinine clearance, TSH, fibrinogen Urine test performed : proteinuria
Blood and urine tests - Year 3 | Year 3
  Description of abnormalities (frequency and percentage) Blood tests performed : lipid profile, glycosylated hemoglobin (HbA1C), cardiac enzymes (troponin C, NT-proBNP), ultra-sensitive C-reactive protein, sodium level, potassium level, urea and creatinine clearance, TSH, fibrinogen Urine test performed : proteinuria
Lying and standing blood pressure tests - Year 3 | Year 3
  Percentage of patients with abnormal blood pressure tests results
Lying and standing blood pressure tests - Year 3 | Year 3
  Description of abnormalities (frequency and percentage)

CONTACTS AND LOCATIONS:
Locations (1):
- Fondation Adolphe de Rothschild, Paris, France

IPD SHARING:
Plan to Share IPD: No